CLINICAL TRIAL: NCT05986955
Title: Food Derived Bacteria and Their Role in Treating Disease
Brief Title: The Impact of Food on Gut Microbiome Composition - a Clinical Trial Determining the Influence of Diet in Gut Microbiome Colonisation and Host Health
Acronym: FIG
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Dr. Sam Forster, Principal Investigator, Monash University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: RES-21-0000-602A
Record Dates: First submitted 2023-07-19; First posted 2023-08-14 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specified Diet 1 - Microbial Diet (Experimental): Participants provided with a typical Australian diet including all food groups as described by the Australian Guide to Healthy Eating without any dietary exclusions. Meals have been designed by researchers and dietitians and prepared by professional chefs.
  Interventions: Other: Diet
- Specified Diet 2 - Non-microbial Diet (Active Comparator): Diet provided to participants is identical to Specified Diet 1 however after cooking and packaging, food for this arm will be sterilised by irradiation in line with International Organisation for Standardisation (ISO) standards and Australian code of good manufacturing practice.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Participants will be assigned prospectively to microbial or non-microbial diet for first phase of trial and will then cross over to the alternate diet following a washout period.

SUMMARY:
The goal of this clinical trial is to examine the impact of food derived bacteria on gut microbiome composition and host health. The main questions it aims to answer are:

* what is the the rate of gastrointestinal colonisation of food derived bacteria?
* what is the contribution of food derived bacteria to gut microbiome stability?

Participants will complete a cross over feeding study of dietitian designed meals of known microbial load and will be asked to provide stool and blood samples for analysis.

DETAILED DESCRIPTION:
To understand the role and stability of food derived bacteria in impacting microbiome composition, 20 healthy participants will be recruited for this single site double blinded randomised controlled crossover pilot trial. The study is divided into four 14 day diet phases - baseline habitual, specified diet 1, habitual washout and specified diet 2. Participants will be randomly assigned to receive a microbial or non-microbial diet in specified diet 1 phase. Each participant will then crossover to receive the alternative diet in the specified diet 2 phase. The microbial and non-microbial diets will be identical except for the removal of naturally occurring food derived bacteria in non-microbial diet. At the commencement of the study and at the end of each diet phase, participants will attend a research clinic to undergo comprehensive clinical and anthropometric assessment and dietary evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Have no genetic conditions (e.g. Prader Willi or Down's Syndrome)
* Not diagnosed with a significant medical conditions (e.g. irritable bowel syndrome, inflammatory bowel disease or type 1/2 diabetes)
* Do not require drug-therapy (e.g. steroids or insulin or antibiotics)
* Not taking dietary supplements, probiotics, prebiotics, symbiotics or fibre supplementation
* Any condition that will affect participation in the study
* Not pregnant, planning a pregnancy or breastfeeding
* Able to complete a two-month dietary study and agree to eating all meals provided
* Have no dietary allergies or dietary restrictions that prevent consumption of provided study meals
* Open bowels regularly - mostly daily
* Able to read, write and understand English

Exclusion Criteria:

* Dietary concerns identified by dietitian
* Aged less than 18 years and older than 65 years
* Diagnosed with a medical condition that requires drug therapy
* Taking medications or supplements known to alter gastrointestinal microbiota
* Women who are pregnant, planning a pregnancy or breastfeeding
* Anyone with a diagnosed gastrointestinal condition/disease e.g. irritable bowel syndrome or inflammatory bowel disease
* Known dietary allergy and/or intolerance, follows a vegan or vegetarian diet, or has coeliac disease
* Anyone with a preference for specific food avoidance or exclusion of certain ingredients in habitual diet
* Unable to tolerate blood collection procedures
* Unable to provide regular stool samples throughout the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Characterisation of gut microbiome | Day 1, 4, 7, 11 and 14 of each phase
  Sequencing and bacterial culturing of stool samples

SECONDARY OUTCOMES:
Participant body mass index (BMI) | BMI will be calculated on day 14 (at end of each diet phase (fortnightly))
  Assessed independently using height and weight measurements and appropriate formula
Participant standing height | Height will be measured on day 14 (at end of each diet phase (fortnightly))
  Measured by stadiometer
Participant weight | Weight will be measured on day 14 (at end of each diet phase (fortnightly))
  Measured using balance scales
Participant waist circumference | Baseline day 1 and end of each 14-day diet phase
  Measured using standard measuring tape
Participant Hip circumference | Baseline day 1 and end of each 14-day diet phase
  Measured using standard measuring tape
Resting systolic and diastolic blood pressure | Blood pressure will be measured on day 14 (at end of each diet phase (fortnightly))
  Measured using digital blood pressure monitor
Mental Health Assessment | Completed at day 1 and end of study (day 56)
  Perceived Stress Scale survey completed by participants
Dietary compliance | Day 1 to Day 14 of specified diet 1 and diet 2 phases
  Measured by participant completed daily diet checklist noting the amount of food they consumed of provided meals during specific diet 1 and 2 phases
Habitual dietary intake | Daily throughout 14-day baseline habitual and habitual washout phases
  Using research food diary mobile phone application
Changes in physical activity levels | Completed at each of each 14-day diet phase
  Using International Physical Activity Questionnaire - Short Form (IPAQ-SF)
Glucose levels | Blood collected at baseline day 1 and day 14 of each phase (fortnightly)
  Blood samples collected will be assessed for glucose levels
Lipid studies | Blood collected at baseline day 1 and day 14 of each phase (fortnightly)
  Blood samples collected will be assessed for lipid studies
Irritable Bowel Syndrome-Severity Scoring System (IBS-SS) | End of each 14-day diet phase
  Completion of Irritable Bowel Syndrome-Severity Scoring System (IBS-SS)
Gastrointestinal symptomatology | Baseline day 1 and day 14 of each diet phase (fortnightly)
  Completion of Gastrointestinal Symptom Rating Scale (GSRS)
Bowel movement | Baseline day 1 and day 14 of each diet phase (fortnightly)
  Completion of Bristol Stool Chart questionnaires
End of study optional semi-structured interview | End of study (at least 8 weeks post-randomisation)
  Interview participants to assess challenges of adhering to study and compliance

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sam Forster, Principal Investigator — Hudson Institue, Monash University
Locations (1):
- BASE Facility, Notting Hill, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Applications made for reasonable access to de-identified study data will be made on a case-by-case basis by the study team. Data-specified appropriate analysis will be determined when required. Applications for data accessibility will be made on a case-by-case basis by study team.
Supporting Information: Study Protocol
Time Frame: Accessibility to individual participant data (IPD) and supporting information will be determined at a later date and on a case-by-case basis
Access Criteria: Accessibility will be assessed on a case-by-case basis